CLINICAL TRIAL: NCT01062451
Title: An ACE Inhibitor or an Angiotensin Receptor Blocker as a Treatment for Methamphetamine Dependence
Brief Title: An ACE Inhibitor (Perindopril) or an Angiotensin Receptor Blocker (Candesartan) as a Treatment for Methamphetamine Dependence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Christopher Verrico, Associate Professor, Psychiatry Research, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: H-23235; R01DA023468 (NIH); DPMC (Other: NIDA); NCT00249665 (obsolete NCT alias)
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Methamphetamine Dependence; Methamphetamine Abuse; Substance Abuse
Keywords: Methamphetamine; Perindopril; Candesartan; Angiotensin receptor blocker; ACE Inhibitor
MeSH Terms: conditions — Substance-Related Disorders | interventions — Perindopril; Sugars; candesartan; candesartan cilexetil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Perindopril (Active Comparator)
  Interventions: Drug: Perindopril
- Candesartan (Active Comparator)
  Interventions: Drug: Candesartan

INTERVENTIONS:
Drug: Perindopril — 8 mg taken orally from days 0 through 7.
  Other Names: Aceon
  Arms: Perindopril
Drug: Placebo — Placebo treatment daily.
  Other Names: Sugar pill
  Arms: Placebo
Drug: Candesartan — 16 mg taken orally from days 0 through 7.
  Other Names: Atacand
  Arms: Candesartan

SUMMARY:
The primary objective is to determine the dose dependent effects of treatment with perindopril on methamphetamine (MA)-induced craving and on the reinforcing effects of MA indexed by MA self-administration. We will also determine the effects of treatment with candesartan on MA-induced craving and on the reinforcing effects of MA indexed by MA self-administration.

DETAILED DESCRIPTION:
Our preliminary data indicate that the ACE inhibitor perindopril can attenuate MA-induced drug craving, suggesting that perindopril should be evaluated as a treatment for MA dependence. Candesartan works similarly to perindopril but should lack the U-shaped dose response. Like perindopril, candesartan is used for hypertension. Whereas perindopril reduces the synthesis of angiotensin II, candesartan blocks angiotensin II receptors.

ELIGIBILITY:
Inclusion Criteria:

* Be English-speaking non-treatment-seeking volunteers.
* Be between 18-55 years of age.
* Meet DSM-IV TR criteria for MA dependence.
* Have a self-reported history of using MA by the IV route.
* Have vital signs as follows: resting pulse between 50 and 90 bpm, blood pressures between 85-150mm Hg systolic and 45-90mm Hg diastolic.
* Have a breathalyzer test indicating an undetectable blood alcohol level upon admission.
* Have hematology and chemistry laboratory tests that are within normal (+/- 10%) limits with the following exceptions: a) liver function tests (total bilirubin, ALT, AST, and alkaline phosphatase) < 3 x the upper limit of normal, and b) kidney function tests (creatinine and BUN) < 2 x the upper limit of normal.
* Have a baseline ECG that demonstrates normal sinus rhythm, normal conduction, and no clinically significant arrhythmias.
* Have a medical history and brief physical examination demonstrating no clinically significant contraindications for study participation, in the judgment of the admitting physician and the principal investigator. Adult ADHD is allowable, as long as symptoms do not interfere with participation.
* Demonstrate MA-induced craving, evidenced by a change in "desire" greater than 20 on a 0 to 100mm VAS.
* Weigh between 60 and 100kg.

Exclusion Criteria:

* Have any previous medically adverse reaction to MA, including loss of consciousness, chest pain, or epileptic seizure.
* Have neurological or psychiatric disorders, such as: episode of major depression within the past 2 years as assessed by MINI; lifetime history of schizophrenia, other psychotic illness, or bipolar illness as assessed by MINI; current organic brain disease or dementia assessed by clinical interview; history of or any current psychiatric disorder which would require ongoing treatment or which would make study compliance difficult; history of suicide attempts within the past three months and/or current suicidal ideation/plan; history of psychosis occurring in the absence of current MA use.
* Meet DSM-IV criteria for abuse or dependence on alcohol or other drugs, except for nicotine or marijuana.
* Have evidence of clinically significant heart disease or hypertension, as determined by the PI.
* Have evidence of untreated or unstable medical illness including: neuroendocrine, autoimmune, renal, hepatic, or active infectious disease.
* Have HIV and are currently symptomatic, have a diagnosis of AIDS, or are receiving antiretroviral medication.
* Be pregnant or nursing. Other females must either be unable to conceive (i.e., surgically sterilized, sterile, or post-menopausal) or be using a reliable form of contraception (e.g., abstinence, birth control pills, intrauterine device, condoms, or spermicide). All females must provide negative pregnancy urine tests before study entry, and weekly throughout the study.
* Have any history of asthma, chronic coughing and wheezing, or other chronic respiratory illnesses.
* Currently use alpha or beta agonists, theophylline, or other sympathomimetics.
* Have any other illness, condition, or use of medications, which in the opinion of the P.I. and/or the admitting physician would preclude safe and/or successful completion of the study.

Rationale for Other Exclusion Criteria:

Participants with asthma or who take medications for asthma are excluded due to potential adverse interactions between treatment medications and MA. Participants who use alcohol heavily are excluded due to the potential of withdrawal symptoms in the hospital. Participants with active HIV disease are excluded to avoid potentially exacerbating their underlying illness and because of potential drug interactions. Reliable methods of birth are required to prevent pregnancy, and the use of frequent urine pregnancy tests will exclude women who become pregnant. This is important because perindopril can produce significant birth defects.

Criteria for Discontinuation Following Initiation:

Participants will be discharged if they have a positive breath test indicating use of alcohol or a urine test indicating use of illicit use of drugs while on the study, if they do not comply with study procedures, or if they do not tolerate MA.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2009-05; Primary Completion 2013-11-20 (Actual); Study Completion 2013-11-20 (Actual)

PRIMARY OUTCOMES:
The dose-dependent effects of an ace inhibitor or an angiotensin receptor blocker on MA- and cue-induced craving and on the reinforcing effects of MA indexed by MA self-administration. | 7 days
  Participants demonstrating MA-induced craving will then be randomized to active study medication (perindopril or candesartan) or matched placebo (day 0). Over days 4 to 7 a variety of procedures will be completed to assess effects of MA and cue-induced craving. On day 7, reinforcing effects will be assessed will be assessed using self-administration procedures.

SECONDARY OUTCOMES:
The effects of an ace inhibitor or an angiotensin receptor blocker on subjective measures. | 7 days
  On days 3 and 5, participants will receive sample doses of 15mg or 30mg MA paired with a dose of placebo saline separated by 180 min, with the order of administration randomized. Subjective effects of MA will be assessed using visual analogue scales (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas F Newton, M.D., Principal Investigator — Baylor College of Medicine
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States